CLINICAL TRIAL: NCT01511640
Title: Behavioral Effects of Drugs (Outpatient)(43)
Brief Title: Behavioral Effects of Pregabalin and Cannabis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Joshua A. Lile, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Joshua A. Lile, Ph.D., Associate Professor of Behavioral Science, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: R01DA036550 (NIH)
Record Dates: First submitted 2012-01-09; First posted 2012-01-18 (Estimated); Results first posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-08

CONDITIONS: Cannabis-use Disorders
Keywords: marijuana; addiction; treatment; pharmacotherapy; cannabinoid
MeSH Terms: conditions — Marijuana Abuse; Behavior, Addictive | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pregabalin 1 (Experimental): Dose 1
  Interventions: Drug: Pregabalin
- Placebo 1 (Placebo Comparator): Placebo 1
  Interventions: Drug: Placebo
- Pregabalin 2 (Experimental): Dose 2
  Interventions: Drug: Pregabalin
- Placebo 2 (Placebo Comparator): Placebo 2
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — pregabalin 2x daily for duration of study
  Arms: Pregabalin 1; Pregabalin 2
Drug: Placebo — placebo 2x daily for duration of study
  Arms: Placebo 1; Placebo 2

SUMMARY:
Cannabis is the most commonly used illicit drug in the United States, and its use is associated with rates of development of abuse and dependence, treatment admission and relapse that are comparable to other illicit drugs. Currently there is no effective pharmacological treatment for cannabis-use disorders. The purpose of the present study is to evaluate the ability of pregabalin to reduce cannabis use thereby evaluating its effectiveness as a medication for cannabis-use disorders.

ELIGIBILITY:
Inclusion Criteria:

* regular cannabis use
* good health other than cannabis use
* willingness to attempt abstinence
* effective form of birth control in female subjects
* available for up to 6 hrs every day for two 2-week test periods with an intervening break of 7-10 days each
* located in close proximity to University of Kentucky

Exclusion Criteria:

* medical screening outcomes outside normal ranges or deemed clinically insignificant
* medical history that would contraindicate pregabalin administration

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua A. Lile, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- Laboratory of Human Behavioral Pharmacology, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 300 mg/Day Pregabalin, Then Placebo: 300 mg/day Pregabalin, then Placebo
  150 mg then 0 mg 2x daily for duration of treatment phase
- Placebo, Then 300 mg/Day Pregabalin: Placebo, then 300 mg/day Pregabalin
  0 mg then 150 mg 2x daily for duration of treatment phase
- 450 mg/Day Pregabalin, Then Placebo: 450 mg/day Pregabalin, then Placebo
  225 mg then 0 mg 2x daily for duration of treatment phase
- Placebo, Then 450 mg/Day Pregabalin: Placebo, then 450 mg/day Pregabalin
  0 mg then 225 mg 2x daily for duration of treatment phase
Period: First Intervention (11-15 Days)
Arm/Group | 300 mg/Day Pregabalin, Then Placebo | Placebo, Then 300 mg/Day Pregabalin | 450 mg/Day Pregabalin, Then Placebo | Placebo, Then 450 mg/Day Pregabalin
Started | 7 | 8 | 7 | 8
Completed | 5 | 8 | 7 | 7
Not Completed | 2 | 0 | 0 | 1
Period: Washout (6-10 Days)
Arm/Group | 300 mg/Day Pregabalin, Then Placebo | Placebo, Then 300 mg/Day Pregabalin | 450 mg/Day Pregabalin, Then Placebo | Placebo, Then 450 mg/Day Pregabalin
Started | 5 | 8 | 7 | 7
Completed | 5 | 8 | 7 | 6
Not Completed | 0 | 0 | 0 | 1
Period: Third Intervention (11-15 Days)
Arm/Group | 300 mg/Day Pregabalin, Then Placebo | Placebo, Then 300 mg/Day Pregabalin | 450 mg/Day Pregabalin, Then Placebo | Placebo, Then 450 mg/Day Pregabalin
Started | 5 | 8 | 7 | 6
Completed | 4 | 7 | 7 | 6
Not Completed | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 300 mg/Day Pregabalin, Then Placebo | Placebo, Then 300 mg/Day Pregabalin | 450 mg/Day Pregabalin, Then Placebo | Placebo, Then 450 mg/Day Pregabalin | Total
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 7 | 8 | 30
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 1 | 5
  Male | 6 | 7 | 5 | 7 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 6 | 8 | 6 | 7 | 27
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 1 | 1 | 6
  White | 6 | 5 | 3 | 7 | 21
  More than one race | 0 | 0 | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Self-administered Puffs of Smoked Cannabis Containing Active THC Concentrations Compared to Placebo Under Controlled Laboratory Conditions
Description: The reinforcing effects of cannabis were determined using a modified progressive ratio procedure in which subjects made 8 choices between puffs of each available cannabis dose and money (US$0.50). The numbered of self-administered puffs of smoked cannabis are measured for each cannabis concentration (0 and 5.9% THC) during active (300 and 450 mg) and placebo (0 mg and 0 mg) pregabalin maintenance.
Time Frame: 9 consecutive choice trials (i.e., no time out between trials) per cannabis dose level.
Measure: Mean (Standard Error); unit: Cannabis puffs
Groups:
- 300 mg/Day Pregabalin: Cannabis choice during 300 mg/day Pregabalin maintenance
  Placebo (0% THC) and Active (5.9% THC) Cannabis
  Pregabalin 300 mg/day
- 0 mg/Day Pregabalin (Placebo 1): Cannabis choice during 0 mg/day Pregabalin maintenance
  Placebo (0% THC) and Active (5.9% THC) Cannabis
  Pregabalin 0 mg/day (comparator for 300 mg/day)
- 450 mg/Day Pregabalin: Cannabis choice during 450 mg/day Pregabalin maintenance
  Placebo (0% THC) and Active (5.9% THC) Cannabis
  Pregabalin 450 mg/day
- 0 mg/Day Pregabalin (Placebo 2): Cannabis choice during 0 mg/day Pregabalin maintenance
  Placebo (0% THC) and Active (5.9% THC) Cannabis
  Pregabalin 0 mg/day (comparator for 450 mg/day)
Arm/Group | 300 mg/Day Pregabalin | 0 mg/Day Pregabalin (Placebo 1) | 450 mg/Day Pregabalin | 0 mg/Day Pregabalin (Placebo 2)
Number analyzed (Participants) | 12 | 12 | 13 | 14
Cannabis puffs
  0% placebo Cannabis | 2.00 (0.92) | 2.67 (0.92) | 3.60 (1.15) | 4.00 (0.88)
  5.9% active Cannabis | 5.75 (0.95) | 5.67 (0.77) | 5.40 (0.85) | 4.80 (0.76)

ADVERSE EVENTS:
Time Frame: 22 days during maintenance on 300 mg pregabalin and matched placebo, and 30 days during maintenance on 450 mg pregabalin and matched placebo.
Groups:
- 300 mg/Day Pregabalin: Cannabis choice during 300 mg/day Pregabalin maintenance
  Placebo (0% THC) and Active (5.9% THC) Cannabis
- 0 mg/Day Pregabalin (Placebo 1): Cannabis choice during 0 mg/day Pregabalin maintenance (placebo comparator for 300 mg/day group)
  Placebo (0% THC) and Active (5.9% THC) Cannabis
- 450 mg/Day PregabalinPregabalin: Cannabis choice during 450 mg/day Pregabalin maintenance
  Placebo (0% THC) and Active (5.9% THC) Cannabis
- 0 mg/Day Pregabalin (Placebo 2): Cannabis choice during 0 mg/day Pregabalin maintenance (placebo comparator for 450 mg/day group)
  Placebo (0% THC) and Active (5.9% THC) Cannabis
Arm/Group | 300 mg/Day Pregabalin | 0 mg/Day Pregabalin (Placebo 1) | 450 mg/Day PregabalinPregabalin | 0 mg/Day Pregabalin (Placebo 2)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13 | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 1/12 | 1/13 | 0/13 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 300 mg/Day Pregabalin (N=12) | 0 mg/Day Pregabalin (Placebo 1) (N=13) | 450 mg/Day PregabalinPregabalin (N=13) | 0 mg/Day Pregabalin (Placebo 2) (N=14)
nausea/vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA | NA — associated with consumption of spoiled food
chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA | NA — associated with injury sustained during excessive use of alcohol

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT01511640/Prot_SAP_000.pdf